CLINICAL TRIAL: NCT05615259
Title: A Prospective, Multi-Center, Randomized Clinical Study of Total Shoulder Arthroplasty Comparing Exactech Guided Personalized Surgery (GPS) vs. Conventional Instrumentation
Brief Title: Comparison Between Exactech Guided Personalized Surgery (GPS) and Conventional Instrumentation of Shoulder Arthroplasty
Status: Recruiting | Type: Observational
Sponsor: Exactech (Industry)
Responsible Party: Sponsor
Other Study IDs: CR18-004
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Technology; Comparison

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to examine the optimization of Reverse Shouder Arthroplasty implant position between GPS and conventional techniques. The secondary objective is to assess the effect of implant position using GPS vs. conventional techniques on ROM and patient reported outcomes. Long-term follow-up to 10 years with minimum 2 year follow-up for patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 21 years of age at the time of surgery
* Patient is indicated for reverse shoulder arthroplasty
* Patient is willing to participate by complying with pre- and postoperative visit requirements
* Patient is willing to participate for the entire length of the prescribed follow-up (minimum 2 years)
* Patient is willing and able to review and sign a study informed consent form
* Preop CT scan is within 3 months of the date of surgery

Exclusion Criteria:

* Revision shoulder arthroplasty
* Reverse shoulder arthroplasty for fracture
* Need for structural glenoid bone graft
* Osteomyelitis of the proximal humerus or scapula; if a systemic infection or a secondary remote infection is suspected or confirmed, implantation should be delayed until infection is resolved
* Inadequate or malformed bone that precludes adequate support or fixation of the prosthesis
* Neuromuscular disorders that do not allow control of the joint
* Significant injury to the brachial plexus
* Non-functional deltoid muscles
* The patient is unwilling or unable to comply with the post-operative care instructions
* Patients who are a known drug or alcohol abuser, or have a psychological disorder (e.g. schizophrenia major depression, bipolar disorder, etc.) as defined by the DSM4 that affect follow-up care or treatment outcomes.
* Alcohol, drug, or other subtance abuse
* Any disease state that could adversaly affect the function or longevity of the implant
* Patient is pregnant
* Patient is a prisoner
* Patient who are currently involved in any personal injury litigation, medical-legal or worker's compensation claims

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet eligibility criteria - Patients who consent to participate to return for follow-up visits out to 10 years
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2020-09-23 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-09-30 (Estimated)

PRIMARY OUTCOMES:
SST-12 | Through study completion, an average of 1 per year
  Shoulder Simple Test (SST) - 12 questions with yes/no responses that measure shoulder pain and function from a patient's perspective - 12 yes corresponds to 100%
SPADI | Through study completion, an average of 1 per year
  Shoulder Pain and Disability Index (SPADI) -13 questions assessing about pain scale (5 questions) and disability scale (8 questions) where 0 indicates no pain/no difficulty and 10 indicates worst pain imaginable/so difficult it requires help while performin these activities
Constant | Through study completion, an average of 1 per year
  Constant Shoulder Score - 100 points scale about pain, Activities of daily living, Strength test, and Range of Motions questions about shoulder where 100 % corresponds to the highest pain
ASES | Through study completion, an average of 1 per year
  American Shoulder and Elbow Surgeons Score (ASES) - 100 points scale about shoulder pain and performance evaluation in activities of daily living where 100 indicates the best shoulder condition
UCLA | Through study completion, an average of 1 per year
  University of California Los Angeles Shoulder Score (UCLA) - 5 Items score which combines both physician (3 items) and patient assessment (2 items) whith a total range from 0-35 where 0 indicates worse shoulder function and 35 better shoulder function outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Hillen, MD, Principal Investigator — Dijklander Ziekenhuis
Locations (1):
- Dijklander Ziekenhuis, Hoorn, Netherlands